CLINICAL TRIAL: NCT01939626
Title: Comparison of Human Embryonic Development Using Sequential and Single Media in IVF Monitored by Time-lapse Imaging.
Brief Title: Comparison of Human Embryo Development Using Sequential and Single Media With Time-lapse Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TL-SCM-2013
Record Dates: First submitted 2013-08-28; First posted 2013-09-11 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Infertility
Keywords: embryo; culture
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: This study was a two-arm, prospective, randomized, controlled clinical trial performed at four independent IVF clinics. Ovarian stimulation and oocyte collection and fertilization were performed as per each clinic's practice. If >6 oocytes from the patient were fertilized, the resulting zygotes underwent stratified randomization into the two different media.
  Allocation was performed in a 1:1 ratio according to a computer-generated randomization list for each couple, which was provided in sealed and numbered envelopes to each clinic.
  Zygotes randomized into G-1/G-2 underwent a media change from G-1 to G-2 on day 3 and subsequent culture until days 5-6. The zygotes randomized to G-TL were cultured continuously without any media change until days 5-6.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To minimize the possible bias for the primary outcome, the embryologist performing the morphologic evaluation on day 3 and 5-6 was blinded to the treatments. The physician, the embryologist, and the couple were also blinded to the culture group from which the embryo had been selected for transfer.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-step medium (Experimental): embryos will be cultured in a single-step medium for 5 days with no change
  Interventions: Device: Single-step medium
- Control (Other): Embryos cultured in two Culture media for 5 Days.
  Interventions: Device: Standard culture medium

INTERVENTIONS:
Device: Single-step medium — This medium will allow in vitro culture of human embryos for 5/6 days
  Other Names: Single step culture medium
  Arms: Single-step medium
Device: Standard culture medium — This culture system needs media change on day 3 of culture.
  Arms: Control

SUMMARY:
The purpose of this study is to compare human embryo in vitro development in sequential and single-step culture medium using time-lapse imaging.

DETAILED DESCRIPTION:
Objective: To study whether a culture medium that allows undisturbed culture supports human embryo development to the blastocyst stage equivalently to a well-established sequential media.

Design: Randomized, double-blinded sibling trial. Setting: Independent in vitro fertilization (IVF) clinics. Patient(s): One hundred twenty-eight patients, with 1,356 zygotes randomized into two study arms.

Intervention(s): Embryos from each patient were randomly allocated into two study arms to compare embryo development on a time-lapse system using a single-step medium or sequential media.

ELIGIBILITY:
Inclusion Criteria:

* 6 or more normal embryos following egg retrieval and fertilization.
* Female patients aged 21-40 years or 21-55 years who are using an egg donor.
* Patients using fresh or frozen ejaculated sperm

Exclusion Criteria:

* Previous history of cancer
* Day 3 embryo transfer

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage of good quality blastocysts | 5 days of in vitro embryo culture
  A cohort of human embryos will be divided into two different media. The ability of the media to support human embryo development will be determined using the standard assessment of the percentage of embryos that achieve a defined embryo grade.

SECONDARY OUTCOMES:
% GQE DAY 3 | Measured 3 days after oocyte pick-up
  Percentage of good quality embryos on day 3 of development
Blast. Utilization rate | Measured 5 and 6 days after oocyte pick-up
  Number of blastocyst that are cryopreserved or transfered on either day 5 or 6 of embryo development.
Blast. rate | Measured 5 and 6 days after oocyte pick-up.
  Number of embryos reaching the blastocyts stage on either day 5 or day 6.

CONTACTS AND LOCATIONS:
Overall Officials: Thorir Hardarson, PhD, Principal Investigator — Fertilitetscentrum AB
Locations (4):
- United States (2):
  - Pacific Fertility Center, San Francisco, California
  - Frisco IVF, Frisco, Texas
- Sweden (2):
  - Fertilitetscentrum, Gothenburg
  - Skanes University Hospital, Malmo

REFERENCES:
- [Derived] Hardarson T, Bungum M, Conaghan J, Meintjes M, Chantilis SJ, Molnar L, Gunnarsson K, Wikland M. Noninferiority, randomized, controlled trial comparing embryo development using media developed for sequential or undisturbed culture in a time-lapse setup. Fertil Steril. 2015 Dec;104(6):1452-9.e1-4. doi: 10.1016/j.fertnstert.2015.08.037. Epub 2015 Sep 25. PMID 26409153